CLINICAL TRIAL: NCT04012411
Title: Study of Brain Derived Neurotrophic Factor (BDNF) Pathway Biomarkers in the Cerebrospinal Fluid in Patients With Huntington's Disease
Brief Title: Study of BDNF Pathway Biomarkers in the Cerebrospinal Fluid in Patients With Huntington's Disease
Acronym: LCR-MH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL19_0081
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Huntington Disease
Keywords: Huntington Disease; CSF; Biomarkers; BDNF; P42
MeSH Terms: conditions — Huntington Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient with LP (Active Comparator): Huntington's disease patients who agreed to have LP
  Interventions: Procedure: Brain MRI; Procedure: Lumbar Punction; Genetic: Blood sample; Other: Cognitive evaluation
- Patient without LP (Active Comparator): Huntington's disease patient with contraindication to LP or refusal to have LP
  Interventions: Procedure: Brain MRI; Genetic: Blood sample; Other: Cognitive evaluation
- Control Group (No Intervention): Retrospective study with biologic samples of patients without Huntington's disease

INTERVENTIONS:
Procedure: Brain MRI — Multimodal brain MRI: volumetry, diffusion tensor, functional rest MRI
  Arms: Patient with LP; Patient without LP
Procedure: Lumbar Punction — Analysis of BDNF, Tau, NFL and TrkB in cerebrospinal fluid
  Arms: Patient with LP
Genetic: Blood sample — Analysis of BDNF, Tau, NFL, and Val66Met polymorphism
  Arms: Patient with LP; Patient without LP
Other: Cognitive evaluation — Symbol Digit Modality Test (SDMT), Stroop test, Trail Making Test, Empan
  Arms: Patient with LP; Patient without LP

SUMMARY:
Huntington disease (HD, 1.3/10 000) is an autosomal dominant disease due to an abnormal expansion of CAG triplets in HTT gene.

Several pathophysiological mechanisms have been evoked, including an alteration of the signaling pathway of the Brain Derived Neurotrophic Factor (BDNF), a neurotrophic factor involved in the survival of neurons (striatal and hippocampal) and synaptic plasticity. BDNF is synthesized at the level of cortical neurons and transported, through the axonal transport in which the Htt is involved, to the nerve endings; it's then secreted in response to excitatory synaptic activity, especially at the level of glutamatergic synapses. Besides, at the postsynaptic level it binds with great specificity to TrkB receptors (tropomyosin-related kinase receptors B) with a neuroprotective effect on dendritic and axonal growth and an increase in synaptic plasticity, especially at the level of the striatum and the hippocampus.

BDNF is decreased in the brain of animal models, as well as in patients with HD; the alteration of this pathway would occur in the early stages of the disease.

In the context of concomitant multiple treatments, the BNDF pathway may be one of the therapeutic targets of HD.

Moreover, in HD it remains essential to detect biological markers representative of the different pathogenic pathways that can be tested in vivo in humans to confirm the hypotheses developed at the level of basic research; these biomarkers could subsequently become biomarkers of disease progression and/or biomarkers of therapeutic efficacy of potential targeted treatments.

Therefore, this study aims to characterize potential biomarkers of the BNDF pathway in plasma and CSF in subjects with HD and to confirm the importance of this pathogenic mechanism in vivo in humans.

DETAILED DESCRIPTION:
* Design: Multicentre prospective case-control study. Centres: University Hospital of Montpellier, France; University Hospital of Bordeaux, France; University Hospital of Nimes, France; University Hospital of Poitiers, France.
* Main objective: To evaluate BDNF in cerebrospinal fluid as a potential marker of the BDNF-TrkB signaling pathway in vivo in HD patients at a symptomatic stage.
* Secondary objectives: i) Evaluate plasma BDNF in subjects with HD; ii) Study the correlation between BDNF in CSF and BDNF in plasma; iii) Study the correlation between markers of the BDNF pathway and clinical severity, multimodal brain MRI parameters, and relevant markers of evolution of HD; iv) Confirm the increase of Tau and NFL (Neurofilament Light Chain) markers in plasma and in CSF, as markers of neuronal degeneration, in subjects with HD ; v) Test the TrkB assay in the CSF of patients with HD
* Inclusion Criteria. General inclusion criteria: age ≥ 18 years old; national health insurance cover. Patient inclusion criteria: genetically confirmed Huntington's disease diagnosis (≥ 35 CAG repeat in HTT gene exon 1); written informed consent; patient agreement for LP, if requested. Control inclusion criteria: previous LP for medical reason; agreement for inclusion in a biobank for research purposes.
* Exclusion Criteria. General exclusion criteria: subject protected by law, under curatorship or guardianship. Patients exclusion criteria: too severe HD, according to the clinician's judgment, possibly making difficult to perform cognitive evaluation or MRI; contraindications to brain MRI; contraindications to LP; inability to give informed consent. Control exclusion criteria: presence of a neurodegenerative of inflammatory central nervous system disease.
* Inclusion period: 48 months
* Duration of participation for each patient: 123 days maximum
* Total research duration: 64 months
* Plan of the study. Patients group: in 90 patients with HD, the investigators will perform: a collection of the main anamnestic and clinical data; a blood test for the determination of plasmatic BDNF, Tau and NFL and the genotyping of the Val66Met polymorphism of the BDNF gene; multimodal brain MRI with volumetry, diffusion tensor, functional MRI of rest; a measurement of the severity of Huntington's disease and Total Functional Capacity scales; neuropsychological tests (SDMT, STROOP test, Trail Making Test (TMT) A and B, digit span). In a subgroup of 45 patients, the investigators will also perform a lumbar puncture for the determination of BDNF, Tau, NFL and TrkB in CSF. Control Group: 45 controls will be selected from the samples present in the existing Biobank with CSF and plasma samples available in Montpellier, France. MRI data will be centralized and processed by the Imaging Institute I2FH Montpellier University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria:

  * age ≥ 18 years-old
  * national health insurance cover
* Patients inclusion criteria:

  * genetically confirmed Huntington's disease diagnosis (≥ 35 CAG repeat in HTT gene exon 1)
  * written informed consent
  * only for patients "with lumbar puncture (LP)": patient agreement for LP
* Control inclusion criteria:

  * anterior LP for medical reason with consent for biobank "Neuro" with following samples present in this biobank : 2 mL blood + 0.5 mL plasma + 0.5 mL cerebrospinal fluid
  * information and non-opposition for the finality of this biobank
  * paired by age with a patient (+/- 5 years difference)

Exclusion Criteria:

* General exclusion criteria:

  * protected by law
* Patients exclusion criteria:

  * Huntington's disease stage too Evolved that may interfere with cognitive evaluations or MRI
  * contraindications to brain MRI
  * only for patients "with LP": contraindications to LP
  * incapacity to give informed consent
* Control exclusion criteria:

  * neurodegenerative of inflammatory central nervous system pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
BDNF(csf) in HD subjects compared to age-matched control subjects (+/- 5 years) | Inclusion
  centralized ELISA assay with Simoa - Quanterix kit technology at the Laboratory of Clinical Proteomic Biochemistry of Montpellier, France.

SECONDARY OUTCOMES:
plasmatic BDNF in HD subjects vs controls | Inclusion
Correlation between BDNF in CSF and BDNF in plasma | Inclusion
Correlation between BDNF and disease parameters | Inclusion
  Correlation between BDNF in CSF or plasma and: disease severity, assessed through a Scale that quantifies the severity of the disease, the disease burden formula [(n.CAG-35.5) x age], the Total Functional Capacity functional scale (TFC), and cognitive scales (Symbol Digit Modalities Test, STROOP test, Trail Making test A and B, direct and indirect digit span); - MRI brain imaging: cerebral and striatal atrophy by morphological imaging, functional resting state MRI, and anatomical connectivity by diffusion tensor imaging
Total Tau and NFL levels in plasma and CSF in HD subjects vs control subjects | Inclusion
TrkBcsf level in subjects with HD vs control subjects | Inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France